CLINICAL TRIAL: NCT01512784
Title: Long Term Immunogenicity of Quadrivalent Human Papillomavirus Vaccine (Gardasil®)in HIV-infected Adolescents and Young Adults vs. Healthy Adolescents and Young Adults: Non-randomized Controlled Clinical Trial
Brief Title: Long Term Immunogenicity of Quadrivalent Human Papillomavirus Vaccine (Gardasil®)in HIV-infected Adolescents and Young Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Gian Vincenzo Zuccotti, Long term Immunogenicity of Quadrivalent Human Papillomavirus vaccine (Gardasil®) in HIV-infected adolescents and young adults vs. healthy adolescents and young adults: non-randomized controlled clinical trial, University of Milan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HLS04/2011
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: HPV; HIV
Keywords: Quadrivalent Human Papillomavirus Vaccine (HPV) Gardasil; HIV infection; Evaluation of quadrivalent HPV vaccine in adolescents and young adults.
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections | interventions — Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

ARMS (2):
- HIV-infected adolescents and young adults (Experimental): female and male HIV-infected subjects aged from 13-27 years old
  Interventions: Biological: Quadrivalent Human Papillomavirus (6, 11, 16 and 18) vaccine (Gardasil ®)
- healthy adolescents and young adults (Active Comparator): female and male healthy adolescents and young adults aged 13-27 years
  Interventions: Biological: Quadrivalent Human Papillomavirus (6, 11, 16 and 18) vaccine (Gardasil ®)

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (6, 11, 16 and 18) vaccine (Gardasil ®) — Human Papillomavirus vaccine (types 6, 11, 16 and 18) (Recombinant, adsorbed).
  Each dose of Gardasil suspension for injection contains 0,5 ml. The shot is usually given in the arm muscle, 3 shots are given on the following schedule:
  First dose: at chosen date. Second dose: 2 months after dose 1. Third dose: 6 months after dose 1.
  Ingredients: highly purified non-infectious protein for each of the Human Papillomavirus types (6, 11, 16 and 18). Each dose (0,5ml) contains approximately:
  Human Papillomavirus type 6 L1 protein 20 micrograms. Human Papillomavirus type 11 L1 protein 40 micrograms. Human Papillomavirus type 16 L1 protein 40 micrograms. Human Papillomavirus type 18 L1 protein 20 micrograms.
  Arms: HIV-infected adolescents and young adults
Biological: Quadrivalent Human Papillomavirus (6, 11, 16 and 18) vaccine (Gardasil ®) — Human Papillomavirus vaccine (types 6, 11, 16 and 18) (Recombinant, adsorbed).
  Each dose of Gardasil suspension for injection contains 0,5 ml. The shot is usually given in the arm muscle, 3 shots are given on the following schedule:
  first dose: at chosen date. Second dose: 2 months after dose 1. Third dose: 6 months after dose 1.
  Ingredients: highly purified non-infectious protein for each of the Human Papillomavirus types (6, 11, 16 and 18). Each dose (0,5ml) contains approximately:
  Human Papillomavirus type 6 L1 protein 20 micrograms. Human Papillomavirus type 11 L1 protein 40 micrograms. Human Papillomavirus type 16 L1 protein 40 micrograms. Human Papillomavirus type 18 L1 protein 20 micrograms.
  Arms: healthy adolescents and young adults

SUMMARY:
Infection with human immunodeficiency virus (HIV) is an important risk factor for HPV infection and the development of HPV-associated lesions in female and male anogenital tract. Data on safety and immunogenicity of quadrivalent human papillomavirus vaccine in HIV-infected population are few. The present study is a non-randomized controlled clinical trial with the primary objective to determine safety ad immunogenicity of quadrivalent human papillomavirus vaccine (Gardasil®) in HIV-infected female and male adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* For both HIV-infected and healthy subjects:

  * Subjects aged 13-27 years, females and males
  * Written informed consent from parent or guardian if applicable (age<18 years)
* For HIV-infected subjects:

  * HIV-positive
  * Asymptomatic subjects (generalized lymphadenopathy is accepted)
  * Lymphocyte CD4+ count > or equal to 350 cells/mm3
* For subjects receiving HAART:

  * Good compliance to therapy
  * At least two suppressed viral loads HIV-RNA (<37copies/ml9 during 6 months prior to enrollment.

Exclusion Criteria:

* For female subjects (both HIV-infected and healthy)
* Pregnancy or breastfeeding
* Total hysterectomy. Participants who have undergone partial hysterectomy and have a cervix are not excluded.
* For both females and males (HIV-infected and healthy):
* Prior vaccination with quadrivalent HPV vaccine Gardasil before study entry.
* History of severe allergic reaction after previous vaccination or hypersensitivity to any vaccine component.
* Any serious chronic or progressive disease (other than HIV) according to the judgment of the investigator:
* Acute infection requiring therapy or fever at time of enrollment
* Chronic autoimmune or oncologic disease receiving chemotherapy
* Concomitant therapies (other than HAART):
* Chronic therapy (for more than 14 days consecutively) with immunosuppressive or immunomodulating agents or chemotherapy during the 6 months prior to study entry.
* Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation prior to study entry.
* Use of investigational agents within 4 weeks prior to study enrollment.
* Current drug or alcohol use or dependence.
* Documented history of non-adherence to antiretroviral treatment regimen within 12 months prior to study entry.

Ages: 13 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
type specific antibody titers for HPV types 6, 11, 16 and 18 at one month after completion of HPV vaccine series (T3) in HIV infected subjects vs. healthy subjects | one month +/- 10 days after 3° vaccine dose
  Immunogenicity of quadrivalent human papillomavirus vaccine (Gardasil®) will be assessed by evaluation of type-specific antibody development for HPV types 6, 11, 16 and 18 from seronegative status at baseline (T0) to seropositive status at one month after the completion of HPV vaccine series (T3), compared with the same immunogenicity testings performed in healthy subjects matched for sex and age.

SECONDARY OUTCOMES:
antibody HPV titers to types 6, 11, 16 and 18, one month after the first two vaccination series (T1 and T2) in HIV-infected subjects vs healthy subjects | one month +/- 10 days after 1°vaccine dose and month+/- 10 days after 2° vaccine dose
  Antibody titers for HPV types 6, 11, 16 and 18 will be evaluated one month after the first (T1) and second (T2) vaccination dose in HIV-infected adolescents and young adults compared with the same immunological testings in healthy adolescents and young adults.
antibody titers to HPV types 6, 11, 16 and 18 at month 12(T4)and 18 (T5)from baseline (T0). | 12 months +/- 10 days and 18 months +/-10 days from baseline
  To assess long-term immunogenicity of quadrivalent human papillomavirus vaccine (Gardasil® in HIV-infected and healthy subjects by evaluation of persistence of HPV antibody titers to types 6, 11, 16 and 18 at month 12 (T4) and 18(T5) from baseline (T0).
local and systemic adverse events | 7 days after each vaccination dose
  Safety and tolerability of three doses of quadrivalent human papillomavirus vaccine (Gardasil ®) in HIV-infected and healthy subjects will be assessed by evaluating the occurrence and severity of local and systemic adverse events during the 7 days after each vaccination dose.
HIV viral load and lymphocyte CD4+ count | baseline (T0), one month after each vaccination dose (T1, T2 and T3) and at month 12 (T4) and 18 (T5) from baseline.
  Longitudinal monitoring of HIV-viral load and lymphocyte CD4+ count will be conducted in HIV-infected subjects from baseline (T0), throughout the study: one month after each vaccination dose (T1, T2, T3) and at month 12 and 18 from baseline (T4, T5).
lymphoproliferative responses, cytokine production and immunophenotype analysis of lymphocyte subpopulations | baseline (T0), one month after 1° vaccination dose (T1) and one month after 3° vaccination dose (T3).
  To evaluate in a subgroup of subjects (20 HIV-infected and 20 healthy) the following immunological parameters at baseline and at 1 month after 1° vaccination dose (T1) and at 1 month after 3° vaccination dose (T3):
  lymphoproliferative responses to HPV-16 L1 from PBMCs in peripheral blood
  Immunophenotype analysis of lymphocyte subpopulations in peripheral blood
  Cytokine production from peripheral lymphocyte subpopulations at baseline and after stimulation with HPV-16 recombinant protein L1.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Vincenzo Zuccotti, Head of Paediatric Department, Principal Investigator — L.Sacco Hospital, via G.B Grassi, 74 20157 Milano, Italy
Locations (1):
- Luigi Sacco Hospital , Department of Paediatrics, via G.B Grassi, 74, Milan, Italy, Italy